CLINICAL TRIAL: NCT03354572
Title: Pilot Study: Postoperative Pain Reduction by Pre Emptive N-Acetylcysteine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maxima Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAC.TEP
Record Dates: First submitted 2017-10-25; First posted 2017-11-28 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study will be a single centre double blinded randomized placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC (Active Comparator): receive 150 mg/kg acetylcysteïne in 200 ml saline (NaCl0,9%) prior to surgery
  Interventions: Drug: Acetyl cysteine
- placebo (Placebo Comparator): receive only NaCl 0.9% prior to surgery (volume identical to active comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Acetyl cysteine — acetyl cysteine 150 mg/kg prior to surgery
  Other Names: NAC
  Arms: NAC
Drug: Placebos — saline 0.9% prior to surgery
  Other Names: Saline 0.9%
  Arms: placebo

SUMMARY:
Despite current available analgesic drugs, post-surgical pain management remains challenging. A potential new target for analgesic drugs are group-II metabotropic glutamate receptors subtypes (mGlu2 and mGlu3 receptors), since growing evidence from animal models show that activation of these receptors produce s analgesic effects in inflammatory and in neuropathic pain states. . N-Acetylcysteine (NAC) is a safe agent and with little to no side effects. NAC can induce analgesia by activating the glutamate:cystein antiporter, causing endogenous activation of the mGlu 2/3 receptors. However, this has only been investigated once in the peri-operative setting, were it showed preliminary promising result of reduction in opiate necessity. In healthy subjects there was a significant reduction in pain ratings to laser stimuli and amplitudes of laser evoked potentials after NAC. Based on these promising results, we hypothesize that pre emptive intravenous NAC can reduce postoperative pain and thereby cause less necessity for escape analgesics like opiates.

DETAILED DESCRIPTION:
Currently approximately 240 million surgical procedures are done worldwide on a yearly basis. lnguinal hernia repair is one of the most performed surgeries in ambulatory setting. Despite currently available analgesic drugs, post surgical pain management remains challenging in this group of patients, as the pain score appears inadequate (mean VAS of 5.8 +/- 1 .22 cm) one day after surgery with the use of common analgesics. Beside accounting for patient discomfort, pain is also a major contributor to prolonged length of hospital stay and is a health care quality indicator. With multimodal pain management the intention is to reduce pain with less side effects of analgesics. Multimodal pain management is the combination of different pharmacologic mechanisms of action, which work by acting at different sites within the central and peripheral nervous system, thereby having an additive or synergistic effect and reducing the necessity of opiates. With this in mind, a potential new target for analgesic drugs are group- ll metabotropic glutamate receptors subtypes (mGlu2 and mGlu3 receptors) localized in the spinal cord and other regions of the nociceptive system. Growing evidence from animal models show that activation of these receptors occur via the glutamate:cystein antiporter and can induce analgesia in models of inflammatory and neuropathic pain. They depress pain transmission at synapses between primary afferent fibers and second order sensory neurons on the dorsal horn of the spinal cord.

N-Acetylcysteine (NAC) is on the market since 1968 and is an over the counter available agent, mostly known for its role as mucolytic agent in cystic fibrosis and for the treatment of acetaminophen intoxication. lt is a safe agent with little to no side effects. Recent studies have shown NAC can inhibit nociceptive transmission in rats and in healthy humans.NAC can induce analgesia by activating the glutamate:cystein antiporter, causing endogenous activation of the mGlu2/3 receptors. Therefore, NAC can potentially become a cheap and safe additive in the multimodal pain management. However, evidence for usage of NAC in the context of multimodal pain management is still lacking. Only one available study in humans evaluated the effect of NAC in the perioperative setting. Despite being a randomised controlled trial, there are several limitations in this study; the study arms are too small and only morphine consumption is presented. Also, blinding might have not as good as suggested since oral NAC has a typical flavour and the placebo was lemonade.

Due to these limitations, still no answer on the question whether NAC can be an additive in current multimodal pain management is provided.

Objective of the study:

Primary Objective:

To evaluate the efficacy of intravenous NAC in comparison with placebo in terms of pain relief after unilateral inguinal hernia repair measured by a visual analogue scale (VAS 0-100) at day 1 after surgery.

Secondary Objective(s):

1. Difference in pain scores between NAC and placebo direct after surgery, before discharge and in following 3 days postoperative.
2. Difference in time before first pain medication is administered postoperative between NAC and placebo.
3. Difference in total consumption of opiates in the hospital (mg) between NAC and placebo.
4. Difference in time from surgery to discharge between NAC and placebo.
5. Difference in postoperative pain medication at home necessary to reach adequate pain relief between NAC and placebo (acetaminophen / NSAID's/ opiates).
6. lf there is a difference in 5, is there also a difference in adverse effects of pain medication (like nausea, obstipation) between NAC and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for laparoscopic unilateral inguinal hernia repair
* ASA 1 or2.
* Age >18 years.

Exclusion Criteria:

* Pregnancy or lactating
* Allergy to NAC
* History of chronic pain
* Use of opioids or neuropathic analgesics
* Use of NAC prior to trial (< 1 month of planned surgery)
* Alcoholism
* Diabetes Mellitus (insulin therapy)
* Asthma or Chronic Obstructive pulmonary Disease
* Known renal function disorders (MDRD <ô0)
* Known liver failure (bilirubin >1.Sx upper limit of normal)
* No written lC by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
pain score day 1 after surgery | 24 hours
  To evaluate the efficacy of intravenous NAC in comparison with placebo in terms of pain relief after laparoscopic inguinal hernia repair measured by a visual analogue scale (VAS 0-100 millimeters) at day 1 after surgery. The higher the score, the more pain the patient has.

SECONDARY OUTCOMES:
direct postoperative pain | <1 hours
  Difference in pain scores between NAC and placebo direct after surgery (1 hour. Measurement in visual analogue scale (VAS 0-100 millimeters) at 1 hour after surgery. The higher the score, the more pain the patient has.
time to first pain medication | <4hours
  Difference in time before first pain medication is administered postoperative between NAC and placebo
total consumption of opiates | <4 hours
  Difference in total consumption of opiates in the hospital (mg) between NAC and placebo
time to discharge | 24 hours
  Difference in time from surgery to discharge between NAC and placebo.
postoperative dosage of analgesics | 72 hours
  Difference in postoperative pain medication at home necessary to reach adequate pain relief between NAC and placebo ( Acetaminophen /NSAID's/opiates).
adverse effects of analgesics | 72 hours
  is there also a difference in adverse effects of pain medication (like nausea, obstipation) between NAC and placebo
Incidence of Treatment-Emergent Adverse Events (e.g. safety of acetylcystein) | <4 hours
  adverse effects of acetylcysteine; do we see exanthema or breathing problems during administration of acetylcystein.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vissers, MD, PhD, Principal Investigator — Chair
Locations (1):
- Maxima Medical Centre, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided, if there is a question for data we will comply as much as possible

REFERENCES:
- [Derived] Mulkens CE, Staatsen M, van Genugten L, Snoeker BAM, Vissers KCP, Bruhn J, Bucx MJL. Postoperative pain reduction by pre-emptive N-acetylcysteine: an exploratory randomized controlled clinical trial. Reg Anesth Pain Med. 2021 Nov;46(11):960-964. doi: 10.1136/rapm-2021-102884. Epub 2021 Aug 26. PMID 34446544

DOCUMENTS (2):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03354572/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03354572/SAP_001.pdf